CLINICAL TRIAL: NCT03020433
Title: Novel Brain Stimulation Therapies in Stroke Guided Expressions of Plasticity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ela B. Plow, Associate Staff, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-128; 16GRNT27720019 (Other Grant/Funding Number: AHA)
Record Dates: First submitted 2016-09-06; First posted 2017-01-13 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Cerebrovascular Disorders; Nervous System Diseases; Brain Diseases; Cardiovascular Diseases; Vascular Diseases; Central Nervous System Diseases
Keywords: Stroke; rehab; rehabilitation; paresis; paralysis; stroke therapy; CVA; cerebrovascular accident; brain diseases; TMS; transcranial magnetic stimulation; CIMT; constraint induced movement therapy; MRI
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Nervous System Diseases; Brain Diseases; Cardiovascular Diseases; Vascular Diseases; Central Nervous System Diseases; Paresis; Paralysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- rTMS Contralesional M1 Inhibition (Active Comparator)
  Interventions: Device: rTMS Contralesional M1
- rTMS Contralesional PMC facilitation (Active Comparator)
  Interventions: Device: rTMS Contralesional PMC
- rTMS Ipsilesional PMC facilitation (Active Comparator)
  Interventions: Device: rTMS Ipsilesional PMC
- rTMS Sham at Ipsilesional M1 (Sham Comparator)
  Interventions: Device: rTMS sham at Ipsilesional M1

INTERVENTIONS:
Device: rTMS Contralesional M1 — 1Hz Contalesional M1 repetitive transcranial magnetic stimulation (1500 pulses, 25 minutes, 90% AMT
  Arms: rTMS Contralesional M1 Inhibition
Device: rTMS Contralesional PMC — 5Hz Contralesional PMC repetitive transcranial magnetic stimulation (1500 pulses, 10 minutes, 5 trains of 300 pulses each with 1 minute rest in between, 90% AMT)
  Arms: rTMS Contralesional PMC facilitation
Device: rTMS Ipsilesional PMC — 5HZ Ipsilesional PMC repetitive transcranial magnetic stimulation (1500 pulses, 10 minutes, 5 trains of 300 pulses each with 1 minute rest in between, 90% AMT)
  Arms: rTMS Ipsilesional PMC facilitation
Device: rTMS sham at Ipsilesional M1 — 1Hz Ipsilesional M1 sham repetitive transcranial magnetic stimulation (1500 pulses, 25 minutes, 50% MSO)
  Arms: rTMS Sham at Ipsilesional M1

SUMMARY:
The investigators ultimate goal is to personalize brain stimulation for stroke so outcomes of the upper limb can be maximized for each individual patient. Several groups including the investigators have recently theorized that personalizing stimulation so as to selectively stimulate iM1 in mild, and cPMd in patients with greater severity would help generalize benefits of stimulation. The investigator premise that variances in expressions of plasticity can explain how to best stratify patients for robust, personalized stimulation.

DETAILED DESCRIPTION:
AIMS: The ultimate goal is to personalize brain stimulation for stroke so outcomes of the upper limb can be maximized for each individual patient. Even though stimulation is one of the most well studied methods to augment plasticity and boost recovery, it is still not approved for outpatient therapy. Benefits of stimulation are weak and variable especially in patients who suffer from greater damage and disability. The key limitation of the standard approach is its generic assumptions about plasticity. The current standard assumes that ipsilesional primary motor cortex (iM1) can impact recovery for patients in all ranges of severity, and intact, contralesional cortices always compete with iM1 to inhibit recovery. But, these long-standing assumptions fail to consider that iM1 or its pathways are damaged in a majority (58-83%) of patients. As such, the potential of iM1 would be weak and variable, and patients will have little option but to rely on plasticity of intact, contralesional cortices that are more likely to survive. Of all surviving cortices, contralesional dorsal premotor cortex (cPMd) expresses plasticity most consistently. cPMd is activated in movement of the paretic limb when activating iM1 is less likely. cPMd even reduces its competition with iM1 and offers its ipsilateral pathways instead to support recovery of the proximal paretic limb when pathways from iM1 are largely damaged.

Several groups including the investigator have recently theorized that personalizing stimulation so as to selectively stimulate iM1 in mild, and cPMd in patients with greater severity would help generalize benefits of stimulation. These theoretical claims, however, remain untested since several gaps exist. For instance, what is the cut-off level of severity that stratifies those who respond to stimulation of iM1 from those who respond to stimulation of cPMd? Even then, are substrates for 'personalized' stimulation same as the substrates that express plasticity in recovery, i.e. if patients benefit from stimulation of cPMd, do they express contralesional plasticity in recovery? Here, the investigator premise that variances in expressions of plasticity can explain how to best stratify patients for robust, personalized stimulation.

ELIGIBILITY:
Inclusion Criteria:

* greater than 21 years old
* more than 6 months from first, unilateral index stroke
* unilateral paresis of the upper limb indexed as greater than or equal to 20% slowness in functional reaching compared to non-paretic limb
* UEFM less than or equal to 61 out of 66.

Exclusion Criteria:

* subjects who cannot perform reaching with shoulder
* severe cognitive deficit (less than or equal to 24 on Mini-Mental State examination.
* contraindication to TMS or MRI including: seizures, ongoing use of certain neuro- or psycho-active medications, implants, or pacemaker.
* currently receiving outpatient therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Aim 1: Change in time (seconds) to perform functional reaching | Change in functional reaching from baseline to post rTMS, assessed for approximately 4-6 hours.
  Patients will be seated with test arm resting on a table. Three buttons (labeled 1, 2, 3) will be arranged in a semi-circle at 80% of reaching distance of the paretic limb. A number (1, 2, or 3) will cue patients to reach and push the designated button as fast as possible using shoulder flexion-abduction and elbow extension while their trunk is stabilized. Three blocks of 20 trials will be tested pre- and post-rTMS.

SECONDARY OUTCOMES:
Aim 2:Change in plasticity evoked with rTMS. | Change in neurophysiology from baseline to post rTMS assessed for approximately 4-6 hours.
  Expressions of plasticity will be noted for ipsilesional vs. contralesional pathways and inhibition imposed on ipsilesional cortices from contralesional cortices. Subjects will be stratified based on which stimulation location evoked the most plasticity from each of the arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ela Plow, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No